CLINICAL TRIAL: NCT05205135
Title: Feasibility Study of Project Carer Matters for Family Caregivers of People With Dementia Receiving Home-based Caregiving
Brief Title: Feasibility Study of Project Carer Matters for Family Caregivers of Persons With Dementia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Geriatric Education and Research Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: GERI1626
Record Dates: First submitted 2021-12-29; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Caregivers; Caregiver Burden; Caregiver Burnout; Dementia
Keywords: Feasibility studies; Caregiver; Nursing; Older person; Singapore
MeSH Terms: conditions — Caregiver Burden; Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Caregivers: Caregivers of persons with dementia supported by the Carer Matters programme
  Interventions: Behavioral: SHARE Programme
- Nurses: Ward nurses who collaborate with the Carer Matters team
  Interventions: Behavioral: SHARE Programme
- Programme facilitators: Facilitators of programmes organised through Carer Matters
  Interventions: Behavioral: SHARE Programme
- Care Support Nurses: Nurses trained to deliver support and assistance as part of Carer Matters Programme
  Interventions: Behavioral: SHARE Programme
- Community partners and hospital leaders: Key policy makers and community leaders who partner with the Carer Matters programme to ensure its success
  Interventions: Behavioral: SHARE Programme
- Other clinicians (e.g. Social workers, Physiotherapists, doctors): Other clinicians who refer caregivers to the Carer Matters programme
  Interventions: Behavioral: SHARE Programme

INTERVENTIONS:
Behavioral: SHARE Programme — SHARE is Singapore's first 'Hospital-to-Home' programme to screen, identify and provide targeted interventions for caregivers at-risk of caregiver burden. Our interventions include psychosocial and emotional preparation of caregivers' mental resilience, and long-term engagement initiatives to connect caregivers into an integrated network of peers and community support services, delivered by programme facilitators and care support nurses.
  Key stakeholders essential for the success of share include ward nurses and clinicians who refer caregivers to SHARE and community partners and hospital leaders.
  This study seeks to recruit all of these individuals to better understand their experience of SHARE and the facilitators and barriers to its successful rollout to better evaluate the feasibility of SHARE in the hospital to home setting.

SUMMARY:
The study uses the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) framework to assess the Carer Matters programme for dementia caregivers in Singapore. A parallel mixed-methods study design is applied to assess the programme's feasibility and effectiveness.

DETAILED DESCRIPTION:
A mixed-methods study to (1) Evaluate the feasibility of Carer Matters for caregivers of PwD and to (2) Explore perspectives of key stakeholders who are directly or indirectly involved with Carer Matters, to better understand the potential sustainability of this framework.

The objectives of are as follows:

1. To explore the perceptions, attitudes and beliefs of family caregivers, healthcare workers and community partners towards Carer Matters.
2. To explore the barriers and facilitators of acceptance and implementation of Carer Matters.
3. To gain insights into the perceived demand of Carer Matters.
4. To gain insights into the family caregivers' preliminary responses to and outcomes from Carer Matters.

The study will involve six inpatient wards of a 1,700-bedded tertiary care hospital which are piloting Carer Matters. These wards comprise of four acute wards and two sub-acute wards. They are selected as they admit a comparatively greater number of patients with dementia than other wards in the hospital. The study will be conducted over 12 months.

Quantitative data is based off programme data collected from all caregivers who undergo Carer Matters. Hence, it will consist of all dementia caregivers whose care recipient is admitted into the pilot wards and agree to participate in Carer Matters.

Qualitative data is based off interviews of key stakeholders of the different components of the Carer Matters programme. The key stakeholders comprises: (1) Family caregivers of PwD (n = 25 to 30), (2) Ward nurses (n= 8 to 10), (3) Care support nurses (n = 2 to 3), (4) Intervention programmes facilitators and standardized patients (n = 3), (5) Community partners and hospital leaders (n = 4), and (6) Other clinicians - medical social workers, physiotherapists, occupational therapists and doctors (n = 4 to 5).

Both qualitative and quantitative data will be triangulated using the RE-AIM framework address the research objectives of the study. These insights will then be used to generate an updated Theory of Change model explaining how SHARE improves caregiver capacity for sustained caregiving. This final model will reflect the processes and mechanisms of Carer Matters that contribute towards the short, medium and long-term outcomes intended, and can serve as a guide for future researchers and practitioners.

ELIGIBILITY:
Inclusion Criteria:

* For family caregivers: (1) Above 21 years of age, (2) The main family caregiver of the PwD receiving home-based care, (3) Able to converse in English language, and (4) Willing to have their interviews audio-recorded.
* For ward nurses: (1) Above 21 years of age, (2) Working as a nurse at one of the inpatient wards piloting SHARE, (3) Referred family caregivers to complete the brief screening tool, and (4) Willing to have their interviews audio-recorded.
* For care support nurses: (1) Above 21 years of age, (2) Involved in either providing direct or indirect patient care to a PwD and their caregiver through SHARE, and (3) Willing to have their interviews audio-recorded.
* For community leaders and hospital leaders: (1) Above 21 years of age, (2) Key decision makers or in leadership positions within the hospital or Working in institutions where there are ongoing or potentially future partnerships with TTSH to provide care services , and (3) Willing to have their interviews audio-recorded.
* For other clinicians: (1) Above 21 years of age, (2) Working as a clinicians at one of the inpatient wards piloting SHARE, (3) Referred family caregivers to complete the brief screening tool, and (4) Willing to have their interviews audio-recorded.

Exclusion Criteria: any potential participant who refuses to have their interviews recorded

-

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible caregivers whose person with dementia are admitted into the pilot wards and receive the SHARE programme will be invited to participate
  All eligible ward nurses and clinicians who work in pilot wards where SHARE is ongoing will be invited to participate.
  All eligible care support nurses and programme facilitators will be invited to participate, as they are all involved in SHARE.
  Eligible hospital leaders and community leaders who have worked with the SHARE programme will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited into programme | Data will be collected over one year, the duration of the first year of the intervention.
  Reach of Carer Matters - Whether Carer Matters Programme affects target population of caregivers. Data collected from programme logs of caregivers recruited not programme and sign-up rates for programmes recommended to participants
Self-reported anxiety scores of CARERS programme participants | Data will be collected over one year, the duration of the first year of the intervention.
  Whether Carer Matters Programme brings about the desired effects in caregiver participants - Reduced anxiety. Data collected through HADS tool administered to caregivers attending CARERS programme.
Self-reported depression scores of CARERS programme participants | Data will be collected over one year, the duration of the first year of the intervention.
  Whether Carer Matters Programme brings about the desired effects in caregiver participants - Reduced depressive symptoms. Data collected through HADS tool administered to caregivers attending CARERS programme.
Self-reported dementia knowledge scores of dementia programme participants | Data will be collected over one year, the duration of the first year of the intervention.
  Whether Carer Matters Programme brings about the desired effects in caregiver participants - Increased dementia knowledge. Data collected through dementia knowledge test designed by team, administered to caregivers attending dementia programme.

CONTACTS AND LOCATIONS:
Overall Officials: Ee Yuee Chan, PhD, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No plans for IPD sharing, due to sensitivity of information shared over interviews.

REFERENCES:
- [Derived] Wu LT, Glass GF Jr, Chew EYH, Ng EJY, Chan EY. Developing a theory of change to guide the design and implementation of a caregiver-centric support service. BMC Health Serv Res. 2024 Dec 18;24(1):1620. doi: 10.1186/s12913-024-11931-y. PMID 39695613
- [Derived] Chan EY, Wu LT, Ng EJY, Glass GF Jr, Tan RHT. Applying the RE-AIM framework to evaluate a holistic caregiver-centric hospital-to-home programme: a feasibility study on Carer Matters. BMC Health Serv Res. 2022 Jul 19;22(1):933. doi: 10.1186/s12913-022-08317-3. PMID 35854296

DOCUMENTS (1):
  • Study Protocol (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT05205135/Prot_000.pdf